CLINICAL TRIAL: NCT05534191
Title: Comparison of Functional and Traditional Strength and Power Training on U19 Soccer Players During Off-season in Norway: A Randomized Controlled Trial
Brief Title: Off-season Training Effects on U19 Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Principal Investigator, Lasse Engberg Treu Lassen, Ph.D. candidate, Aalborg University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 438956
Record Dates: First submitted 2022-08-26; First posted 2022-09-09 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Soccer Performance
Keywords: Technical skills; Power; Coordination; Speed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention (Experimental): This group will use a functional training system developed specifically for football players to improve their physical strength and movement abilities on the field.
  Interventions: Other: Experimental, comparator and control
- Positive control (Active Comparator): This group will use general strength exercises with the purpose of improving physical strength.
  Interventions: Other: Experimental, comparator and control
- Negative control (No Intervention): Control group A group that is not treated

INTERVENTIONS:
Other: Experimental, comparator and control — To quantify the effect of a strength intervention for footballers on improved range of motion, balance, speed, jump height, and technical football skills compared to a training group performing basic power exercises and machine-based strength training and a control group.
  Arms: Intervention; Positive control

SUMMARY:
The goal of this randomized controlled trial is to evaluate whether functional strength and power training or traditional strength and power training during the off-season can improve soccer-specific performance in trained male U19 Norwegian soccer players.

The main questions it aims to answer are:

Does functional training lead to greater improvements in technical soccer skills (passing, shooting, dribbling) compared to traditional training?

Do both training modalities improve mobility, dynamic balance, sprint speed, change of direction, and jumping performance?

Researchers will compare the functional training group, the traditional training group, and a control group to see if either training approach provides superior performance benefits.

Participants will:

Take part in an 8-week intervention.

Complete two weekly strength sessions (functional or traditional depending on allocation).

Attend two weekly soccer sessions during the first 4 weeks (all groups).

Undergo a standardized test battery measuring mobility, balance, technical skills, sprinting, change of direction, and vertical jump before and after the intervention.

ELIGIBILITY:
Inclusion Criteria

Male soccer players aged 16-20 years.

Active competitors in the Norwegian G19 0. Division or the Norwegian Tipping League (Senior 3. Division).

Minimum of eight years of organized soccer experience.

At least two years of structured resistance training experience.

No concurrent involvement in other structured physical activity programs.

Exclusion Criteria

History of lower-limb injury within the past three months.

Inability to meet the required training attendance (≥14 out of 16 sessions).

Participation in additional structured training programs outside the intervention.

Ages: 16 Years to 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 53 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-01-14 (Actual); Study Completion 2024-01-14 (Actual)

PRIMARY OUTCOMES:
Loughborough soccer passing test | Day 1
  Measure precision in passing (Seconds)
Loughborough soccer passing test | 2 months
  Measure precision in passing (Seconds)
Loughborough soccer shooting test | Day 1
  Measure precision in shooting and reaction (Points and secounds )
Loughborough soccer shooting test | 2 months
  Measure precision in shooting and reaction (Points and secounds )
Agility with ball | Day 1
  Measure technical abilities with the ball (Seconds)
Agility with ball | 2 months
  Measure technical abilities with the ball (Seconds)

SECONDARY OUTCOMES:
Active knee extension test | Day 1
  Measure range of motion (Degrees)
Active knee extension test | 2 months
  Measure range of motion (Degrees)
Hip External rotation | Day 1
  Measure range of motion (Degrees)
Hip External rotation | 2 months
  Measure range of motion (Degrees)
Hip Internal rotation | Day 1
  Measure range of motion (Degrees)
Hip Internal rotation | 2 months
  Measure range of motion (Degrees)
Active dorsi flexion test | Day 1
  Measure range of motion (Degrees)
Active dorsi flexion test | 2 months
  Measure range of motion (Degrees)
Dynamic leap balance test | Day 1
  Measure improved dynamic balance (Secounds)
Dynamic leap balance test | 2 months
  Measure improved dynamic balance (Secounds)
S180 sprinting test | Day 1
  Measure change of direction abilities (Secounds)
S180 sprinting test | 2 months
  Measure change of direction abilities (Secounds)
Vertical jumping test | Day 1
  Measure jumping abilities (Cm)
Vertical jumping test | 2 months
  Measure jumping abilities (Cm)
10 m and 20 m linear sprint | Day 1
  Measure the ability to accelerate and maximum speed (Seconds; Km/h)
10 m and 20 m linear sprint | 2 months
  Measure the ability to accelerate and maximum speed (Seconds; Km/h)

CONTACTS AND LOCATIONS:
Locations (1):
- SSA Steinkjer, Steinkjer, Trøndelag, Norway